CLINICAL TRIAL: NCT00631748
Title: A Double-Blind, Placebo-Controlled Trial of the Efficacy of Quetiapine for the Reduction of Cocaine Use
Brief Title: Quetiapine for the Reduction of Cocaine Use
Acronym: AZC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA1 42; IRUSQUET0449 (Other Grant/Funding Number: Astra/Zeneca Pharmaceuticals)
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Cocaine Dependence; Cocaine Abuse; Cocaine Addiction; Drug Abuse; Substance Abuse
Keywords: cocaine; quetiapine fumarate; dependence; abuse; addiction; treatment
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Quetiapine Fumarate; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Drug (Experimental): Subjects randomized to the experimental arm of the study will be initially administered 50mg/day quetiapine fumarate (Seroquel XR) to be titrated up to 400mg/day by the end of the second week. Subjects will be stabilized at a dose of 400mg/day or alternatively 300, 200, 100, or 50mg/day or quetiapine fumarate as tolerated. During the 12 week treatment phase, all subjects attended weekly group cognitive-behavioral therapy sessions. This therapy platform utilized the cognitive-behavioral therapy manual, Seeking Safety. Seeking Safety has been shown to effectively reduce substance use and to improve psychological functioning in a variety of populations.
  Interventions: Drug: quetiapine fumarate; Behavioral: Cognitive-behavioral Therapy
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm of the study will follow the same titration and dosing procedure as the experimental arm but will receive matched placebo tablets. During the 12 week treatment phase, all subjects attended weekly group cognitive-behavioral therapy sessions. This therapy platform utilized the cognitive-behavioral therapy manual, Seeking Safety. Seeking Safety has been shown to effectively reduce substance use and to improve psychological functioning in a variety of populations.
  Interventions: Drug: Matched Placebo; Behavioral: Cognitive-behavioral Therapy

INTERVENTIONS:
Drug: quetiapine fumarate — At baseline, subjects in the experimental group will initially be administered 50 mg/day of Seroquel XR™ (extended release formulation of quetiapine fumarate), to be titrated up to 400 mg/day of Seroquel XR™ by the end of the second week. By the end of week 2, subjects will be stabilized on a dose of 400 mg/day or alternatively 300, 200, 100, or 50 mg/day of study drug, as tolerated. If a subject is unable to tolerate the 50 mg/day dose, he or she will be discontinued from the drug portion of the study.
  Other Names: Seroquel XR
  Arms: Study Drug
Drug: Matched Placebo — Subjects randomized to the placebo comparator group will follow the same titration and dosing procedures as the experimental group, but will receive matched placebo tablets.
  Arms: Placebo
Behavioral: Cognitive-behavioral Therapy — During the 12 week treatment phase, all subjects attended weekly group cognitive-behavioral therapy sessions. This therapy platform utilized the cognitive-behavioral therapy manual, Seeking Safety. Seeking Safety has been shown to effectively reduce substance use and to improve psychological functioning in a variety of populations.

SUMMARY:
This placebo-controlled trial will test the effectiveness of Seroquel XR™ for the treatment of cocaine dependence in non-psychotic individuals who are cocaine dependent.

DETAILED DESCRIPTION:
Cocaine abuse continues to be an epidemic. Co-morbid psychiatric disorders and high risks behaviors compound the morbidity, economic costs, and social destruction associated with this public health crisis. This is a 12 week, prospective, intent-to-treat, double-blind, randomized, placebo-controlled study of Seroquel XR™ versus matched placebo, combined with cognitive-behavioral group therapy, for the treatment of cocaine dependence in non-psychotic individuals.

We will conduct this study at the American Lake (Tacoma) and Seattle campuses of the VA Puget Sound Health Care System, recruiting veteran and non-veteran participants currently using cocaine from the greater Pierce and King Counties region. It is anticipated that 120 subjects will be consented and screened for study participation and that 60 subjects will be randomized to treatment.

After subjects have provided informed consent, they will enter a 1 week screening phase during which medical, psychiatric, and substance use measures and assessments will be administered to determine study eligibility. At baseline, we will assess cocaine use, cocaine craving, psychiatric symptoms, and high risk behaviors. Also at this visit, subjects will be randomly assigned to treatment with quetiapine (target dose 400 mg/day) or placebo. During the treatment phase, subjects will visit the clinic once a week for safety monitoring, completion of ratings and questionnaires, UDS's, and participation in a cognitive-behavioral therapy group. At end of study, week 12, a physical examination will be administered and a UDS and clinical laboratory values obtained. In addition, substance use, psychiatric symptoms, and high risk behaviors will be assessed. To monitor safety and further evaluate treatment effects, we will ask participants to return for a follow-up visit at week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Males and females aged 18-65 years
3. Female subjects of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at the screening and baseline visits and agree to use one of the following methods of birth control: a) oral contraceptive, b) patch, c) intrauterine progesterone or non-hormonal contraceptive system, d) levonorgestrel implant, e) medroxyprogesterone acetate contraceptive injection, or f) complete abstinence from sexual intercourse
4. A diagnosis of current cocaine dependence; as determined by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders 69 (SCID-I/P)
5. Has used cocaine within the 30 days prior to screening
6. Able to understand and comply with the requirements of the study
7. Is seeking treatment for cocaine dependence
8. Is able to provide a reliable primary contact phone number and is able to provide a reliable alternate contact address and phone number, such as for a relative or close friend
9. Anticipates no life changes that would preclude study completion

Exclusion Criteria:

1. Pregnancy or lactation
2. Currently hospitalized or in a detoxification program
3. Physiological dependence on alcohol, sedative/hypnotic, or any other substance requiring medical detoxification
4. Current diagnosis of psychotic disorder, including bipolar disorder with psychotic features, as determined by the SCID-I/P or clinical interview
5. Subjects who are judged by the investigator to be psychiatrically unstable, including posing an imminent risk of suicide or a danger to self or others, as determined by the SCID-I/P, CGI-S, Hamilton Anxiety Rating Scale(HAM-A), Hamilton Rating Scale for Depression(HAM-D), or clinical interview
6. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
7. Has a history of neuroleptic malignant syndrome or other serious adverse reaction to antipsychotic medication
8. Use of any antipsychotic medication within the 30 days preceding baseline
9. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days prior to baseline including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluoxetine, fluvoxamine, paroxetine, and saquinavir
10. Use of any of the following cytochrome P450 inducers in the 14 days prior to baseline including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
11. Evidence of any clinically relevant disease (e.g., renal, hepatic, gastrointestinal, pulmonary, cardiac, or cerebrovascular disease, AIDS, cancer, asthma, neurological or neuromuscular disease, seizure disorder, or clinically significant abnormal laboratory value) or any clinical finding that in the judgment of the investigator could potentially be negatively affected by study participation or that could potentially affect study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Tapp, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Tacoma, Washington, United States

REFERENCES:
- [Background] Kennedy A, Wood AE, Saxon AJ, Malte C, Harvey M, Jurik J, Kilzieh N, Lofgreen C, Tapp A. Quetiapine for the treatment of cocaine dependence: an open-label trial. J Clin Psychopharmacol. 2008 Apr;28(2):221-4. doi: 10.1097/JCP.0b013e318166f50d. PMID 18344735
- See also: Website for Seeking Safety — http://www.seekingsafety.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of cocaine dependence were recruited from the VA Puget Sound Health Care System and the local community.
Pre-assignment Details: A screening visit was conducted to ensure that they met inclusion/exclusion criteria for the study. If they met criteria, they were scheduled for a baseline visit, during which they were randomized to either the quetiapine or placebo arm of the study.
Groups:
- Study Drug: Oral quetiapine
- Placebo: Placebo (sugar pill)
Period: Overall Study
Arm/Group | Study Drug | Placebo
Started | 29 | 31
Completed | 11 (11 participants completed the double-blind portion of the study; 8 participants completed follow-up.) | 9 (9 participants completed the double-blind portion of the study; 5 participants completed follow-up.)
Not Completed | 18 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.11 (6.97) | 47.71 (9.69) | 47.90 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 26 | 26 | 52
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Timeline Followback Interview (TLFB)
Description: The primary outcome measure was the self-report of cocaine use in the past week, as assessed with a Timeline Followback Interview (TLFB). The TLFB is a questionnaire in which the subject is asked to self-report how much cocaine was used and how much money was spent on cocaine every day for the past 1-2 weeks.
Time Frame: Grams of cocaine used at end of study (12-weeks)
Population: At end of study(12-weeks) 11 participants remained in the quetiapine group and 9 participants remained in the placebo group.
Measure: Mean (Standard Deviation); unit: grams of cocaine used
Groups:
- Study Drug: Quetiapine (Seroquel XR)
- Placebo: matched placebo (sugar pill)
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 11 | 9
grams of cocaine used | 0.11 (0.30) | 0.63 (1.78)
Statistical Analysis 1: Comparison: Study Drug vs Placebo; We used a repeated-measures ANCOVA to compare cocaine usage between the two groups. This incorporated the multiple administrations of the Timeline Followback measure; Test type: Superiority or Other; p < 0.25, ANCOVA; We compared TLFB at baseline and at end of study

2. Secondary Outcome: Percentage of Participants Attaining Abstinence for Three Weeks
Description: Abstinence was defined as a negative urine drug screen (UDS) (for cocaine) for three consecutive weeks of the trial measure at either time point Week 6 or Week 12
Time Frame: Abstinence defined as negative UDS for 3 consecutive weeks of the trial
Population: At end of study (12-weeks) 11 participants remained in the quetiapine group and 9 participants remained in the placebo group.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: match placebo (sugar pill)
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 11 | 9
Percentage of Participants | 45.5 | 44.4
Statistical Analysis 1: Comparison: Study Drug vs Placebo; End-of-trial abstinence was defined as a negative urine drug screen (for cocaine) for three consecutive weeks at the end of the study; Test type: Superiority or Other; p = .65, Regression, Cox

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire time the subject was enrolled in the study, including the screening, 12-week clinical trial, and 4 week follow-up appointment.
Arm/Group | Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/31
Other Adverse Events (participants affected / at risk) | 22/29 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=29) | Placebo (N=31)
Respitory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Subject was in quetiapine arm, but was not taking the study medication at the time of the adverse event, which appeared related to cocaine use and subsequent secondary infection.
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=29) | Placebo (N=31)
Akathesia (Psychiatric disorders) | 9 (10) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Dizziness/Lightheadedness (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Drowsiness/Hypersomnia (General disorders) | 17 (17) | 10 (10)
Dry Mouth (General disorders) | 17 (17) | 6 (6)
Heartburn (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 3 (3)
Increased Appetitie (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Insomnia (General disorders) | 10 (10) | 11 (11)
Menstral Irregularities (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Orthostasis (Vascular disorders) | 5 (5) | 4 (4)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Urinary Hesitancy (Renal and urinary disorders) | 3 (3) | 3 (3)
Weight Gain (General disorders) | 8 (8) | 2 (2)
Sexual Dysfunction (Reproductive system and breast disorders) | 8 (8) | 4 (4)

LIMITATIONS AND CAVEATS:
1) High number of drop-outs (68%) means that analyses are limited by a lack of power. 2) More males than females included-may reflect differences in cocaine drug usage between the sexes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No